CLINICAL TRIAL: NCT06538506
Title: ANIMATOR - A Single-blind Randomized Controlled Trial of RehUP BCI Controlled Robotic Therapy vs. an Attention-based Control
Brief Title: ANIMATOR - RehUP BCI Controlled Robotic Therapy vs. an Attention-based Control
Acronym: ANIMATOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: VIBRAINT Inc. (Unknown)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANIMATOR
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Stroke
Keywords: Brain Computer Interface; Robotic Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups for the duration of the study (BCI therapy or standard physiotherapy employing active and passive range of motion exercises).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessor and investigator will be blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RehUp BCI intervention (Experimental): The BCI intervention will complete 24 one hour intervention sessions (3x/week for 8 weeks).
  Interventions: Device: RehUp BCI Intervention
- Control Therapy (Active Comparator): Participants randomly allocated to the control therapy arm will complete 24 one hour therapy sessions (3x/week for 8 weeks).
  Interventions: Other: Control Therapy

INTERVENTIONS:
Device: RehUp BCI Intervention — Participants will be seated wearing a cap on their head containing surface electrodes connected to a computer/laptop. The laptop employs machine learning algorithms and uses the scalp electroencephalogram (EEG) signals from the scalp's surface to control a robotic arm which supports the patient's stroke-affected arm. The machine learning algorithms rapidly interpret EEG signals and adjust the outgoing movement commands to the robot based on an individual's responses to stimuli. The participant will be wearing a VR headset. The VR displays visual stimulus in time with the robotic arm. Based on information from the EEG, the participant is able to animate their robotic arm and receive visual task-based feedback in the VR.
  Arms: RehUp BCI intervention
Other: Control Therapy — The study therapist will focus on 3 activities (~15 minutes each/session): passive range of motion exercises, motor imagery, and mirror therapy. These activities were chosen as they are all passive activities that are commonly used in a patient with severe impairment of the post-stroke arm and hand. Each session will last ~1hour including set up and switching between activities.
  Arms: Control Therapy

SUMMARY:
ANIMATOR aims to examine how BCI therapy vs. attention based control therapy can be used to treat people in the chronic phase of stroke with moderate to severe upper extremity impairment. This interventional trial has two phases: Pilot (10 consecutive days of intervention) and a Randomized Phase (24 sessions over 8 weeks).

DETAILED DESCRIPTION:
There is a large population of Canadians with chronic stroke and severely impaired upper limbs. Consultation with this population reveals individuals who are looking for treatment to improve their ability to move their arm and hand. The aim of the trial is to offer such a post-stroke neurorehabilitation solution using the RehUp brain computer interface (BCI). To do so, the investigators will harness neuroplastic mechanisms that form new connections in the brain helping the participant to move their arm and hand voluntarily outside of BCI and robotic support.

Given the potential for BCI facilitated post-stroke therapy to improve upper extremity function, the investigators will conduct a pilot trial and then a randomized controlled trial to compare the responses of the upper extremity in chronic stroke survivors to RehUp BCI controlled robotic device vs. an attention-based control comparator.

ANIMATOR is a phase 2, prospective, open label, randomized, controlled trial with blinded outcome assessment. Randomization will be centrally blocked and computerized. Participants will be randomized 1:1 BCI intervention or control.

In the Pilot phase, 10 participants will be enrolled and all allocated to the intervention arm.

In the Randomized Phase, Forty stroke survivors more than 6 months post-stroke with severe arm impairment will be recruited for this trial. Participants will complete 24 one-hour sessions (3x/wk for 8 weeks) of BCI robotic upper extremity therapy, or a control intervention. Potential participants will be identified by stroke physiatrists, neurologists and therapists working in clinics with individuals with stroke related impairment. They may also be identified through previous participation in research studies at one of the trial sites or through self-identification in response to community outreach by the investigators to local stroke recovery groups. Consent will be acquired prior to participating in the study. Participant will be screened using the Fugl-Meyer Upper Extremity (FM-UE), Modified Ashworth Scale (MAS), and Visual Acuity measures to meet inclusion criteria after they have consented to participate.

All groups will receive standard of care rehabilitation. Participants will not be blinded, but the assessor therapist will be. These therapists will complete a training session with the central site to ensure replicability between sites and assessors. Blinded assessors will never deliver either intervention in the trail.

The BCI intervention uses the VIBRAINT BCI robot. It allows participants to perform tasks in a virtual reality environment. In the VR,the participant is given a task to either focus on the motor goal (a target virtual object) or imagine motion of the paralyzed arm connected to this object while reaching to it or grasping it. Once the BCI recognizes cortical activity related to the assigned task, it sends a message to the robotic device to accomplish the desired motion, complemented by synchronous movement in Virtual Reality (VR) of the participant's avatar's arm. During the robotic-driven motion the participant imagines the movement as if it is being performed by them voluntarily. The participant will perform a series of tasks in VR focused on improving arm and hand function. These tasks will be scaled in difficulty and tailored to the participant's level of impairment. The goal is for the participant to complete as many repetitions as possible. A therapist will supervise these sessions to ensure the participant does not become too fatigued. The session will last 45 minutes.

The control intervention is completed with a therapist and focuses on three activities: passive range of motion exercises, motor imagery, and mirror therapy for 15 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors, ≥ 6 months post-stroke with severe arm impairment.
* 18 years of age of older
* Adequate language skills to be able to follow instructions
* FM-UE score 30 or less at study entry (i.e., severe arm impairment and would likely not use the stroke-affected arm in daily activities)
* Modified Ashworth Score ≦ 2
* Visual acuity 20/50 corrected (both eyes)

Exclusion Criteria:

Potential participants will be excluded if they do not meet the requirements above, or:

* have neurologic history in addition to stroke (injury or disease), eg. TBI, MS, dementia
* enrollment in concurrent interventional trial
* major co-morbid illness making study completion unlikely
* contraindication to MRI (such as pacemaker, pregnancy, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity (FM-UE) | Baseline, 4weeks, 8 weeks, 16 weeks
  Change in Fugl-Meyer Upper Extremity (FM-UE) from measurement at baseline. The FM-UE is the most widely used outcome measure for upper limb stroke recovery studies.
  The FM-UE is scored on a scale from 0 to 66, where 66 points indicates unimpaired motor function.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in Action Research Arm Test (ARAT) from measurement at baseline. The ARAT will provide complimentary data on limb impairment.
  The ARAT is scored on a scale from 0 to 57 points, where 57 points indicates unimpaired motor function.
Modified Ashworth Scale (MAS) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in Modified Ashworth Scale (MAS) from measurement at baseline. The MAS is used to assess spasticity.
  The MAS is scored on a 6 point scale [0, 1, 1+, 2, 3, 4]. 0 indicates no increase in tone. 4 indicates the limb is rigid in flexion or extension.
Patient Health Questionnaire - Module 9 (PHQ-9) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in Patient Health Questionnaire - Module 9 (PHQ-9) from measurement at baseline. The PHQ-9 is used to screen for depression.
  The PHQ-9 is a 10 question screening tool where nine of the ten items are scored on a scale from 0 to 3. The tenth item grades how difficult the first nine items make the participant's day-to-day life. A lower score indicates a lower likelihood and/or severity of depression.
EQ-5D (EuroQuol Measure of Health Status, Version 5D) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in EQ-5D (EuroQuol Measure of Health Status, Version 5D) from measurement at baseline. The EQ-5D is used to measure quality of life.
  The EQ-5D scores fives areas of health on a scale of 1-5, where 1 indicates no problems and 5 indicates extreme problems.

OTHER OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in National Institute of Health Stroke Scale (NIHSS) from measurement at baseline. The NIHSS is used to measure stroke severity.
  The NIHSS evaluates 11 items on 3, 4, or 5 point scales depending on level of detail. Higher scores indicate more severe symptoms of stroke.
Modified Rankin Scale (mRS) | Baseline, 4 weeks, 8 weeks, 16 weeks
  Change in Modified Rankin Scale (mRS) from measurement at baseline. The mRS is used to measure the degree of functional neurological disability after stroke.
  The mRS is a 7 point scale (0-6) where 6 indicates that the patient has died and 0 indicates the patient has no symptoms of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Dukelow, MD PhD FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers.